CLINICAL TRIAL: NCT05041465
Title: The Cosmetic Effect of Mineral Clay Masks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1296789
Record Dates: First submitted 2021-03-05; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Rhytides

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- French Green Clay Mask (Experimental)
  Interventions: Other: Clay mask
- Rhassoul Clay Mask (Experimental)
  Interventions: Other: Clay mask
- Bentonite Clay Mask (Experimental)
  Interventions: Other: Clay mask

INTERVENTIONS:
Other: Clay mask — Clay mask powders- French green, Rhassul and bentonite

SUMMARY:
The aim of this study is to evaluate the cosmetic effects of commercially available mineral clay masks over a 4-week period. Changes in skin pigmentation, shine, wrinkles, and texture will be assessed.

A second aim of the study is to assess the safety and tolerability of mineral clay masks by assessing redness and participant feedback.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-50
* Individuals in good general health
* Individuals free of any autoimmune or systemic disorder, which would interfere with the analysis.

Exclusion Criteria:

* Individuals who have been on any topical prescribed medications for the past 2 weeks
* Individuals who have history of acute or chronic disease that would likely interfere with or increase the risk on study participation at the discretion of the investigator
* Individuals with active (flaring) disease or chronic skin allergies (atopic dermatitis/eczema) or those who have recently undergone treatment for skin cancer (within the last 12 months) in the area of testing on the forehead, nose and the cheeks
* Female volunteers who are pregnant or planning to become pregnant over the course of the study. The risk to pregnant women is minimal but the facial appearance can be confounded by the altered hormones associated with pregnancy, as is well documented in chloasma which is dyspigmentation that arises in pregnancy. Women who become pregnant during the duration of the study will become ineligible but there are no birth control requirements.
* Female volunteers who have started a new hormonal birth control agent or switched to a hormonal birth control agent within the past 60 days
* Individuals who have had any medical or cosmetic procedure, such as laser resurfacing, or plastic surgery to the test site (face) within the last 6 months. This includes botulinum toxin, dermal fillers, collagen or other similar cosmetic procedure
* Individuals who are currently using or during the past 14 days have used a retinoid such as tretinoin, adapalene, or retinol containing agents or a hydroquinone containing agent
* Individuals who have used mineral clay masks on their face within the last 14 days
* Individuals with a known history of hypersensitivity to any ingredients to the agent that is being assessed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Count of Participants with Decrease in Skin pigmentation intensity at 4 Weeks | 4 weeks
  Computer and photography based facial image analysis

SECONDARY OUTCOMES:
% of Participants with Skin redness intensity improvement at 4 weeks | 4 weeks
  Computer and photography based facial image analysis

OTHER OUTCOMES:
Patient tolerability survey | 4 weeks
  Survey to grade for side effects

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided